CLINICAL TRIAL: NCT05948514
Title: Venous Thromboembolism and Infections Associated With Three Vascular Access Devices in Home Parenteral Nutrition : a Prospective Cohort Study
Brief Title: Complications Related to Vascular Access Devices in Home Parenteral Nutrition Patients
Acronym: CRVADHPNP
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL22_1128
Record Dates: First submitted 2023-07-05; First posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Vascular Access Complication
Keywords: central venous access device; catheter-related complications; venous thromboembolism; catheter-related bloodstream infection; peripherally inserted central catheters; home parenteral nutrition
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- adult patients followed up in the nutrition and access device was inserted for parenteral nutrition: no intervention, observational study patients are enrolled, and followed up until a catheter related complication occurs
  Interventions: Other: The complications related to central venous access device

INTERVENTIONS:
Other: The complications related to central venous access device — The complications related to central venous access device were collected when occurs : from time of catheter insertion, until first complication, or removal for another type of catheter, or until death.

SUMMARY:
Central vascular access devices are required for home parenteral nutrition (HPN). There is few data available concerning their complications in adult HPN patients, and the potential link between venous thromboembolism and catheter infection is not well established.

The aim of this prospective cohort study is to compare the incidence rate of catheter related complications among 3 types of central vascular access: peripherally inserted central catheters; tunneled catheters and port-a-cath devices, in adults patients on HPN; describe the risk factors, and identify a potential link between venous thromboembolism and infection.

More than 300 patients will be consecutively enrolled and followed up from the time of catheter insertion until its removal. Venous complication (identify by an ultrasound examination if deep vein thrombosis is suspected), infection related to catheter and mechanical complications will be analyzed. The incidence of complications will be expressed per 1000 catheters-day and or as a percentage of total catheter.

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* having a catheter insertion during the study periode
* at the unit of vascular access of Lyon Sud Hospital
* for parenteral nutrition
* from July 1st, 2017 to June 30, 2020

Exclusion Criteria:

* catheter inserted in intensive care unit
* for other treatment (chemotherapy, antibiotic)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients receiving HPN
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Rate of (incidence) symptomatic venous thromboembolism, catheter related infection, and mechanical complications related to central venous access device | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  * Deep vein thrombosis of the upper extremity : suspected if symptomatic (swelling, local pain, edema) and confirmed by venous ultrasound and/or computed tomography
  * Catheter related bloodstream infection suspected if local inflammation and/or fever, and confirmed by blood sample and/or catheter culture
  * Mechanical complications (displacement, drop, kink) : described by nurses or patient

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Lyon Sud-Hospices Civils de Lyon, Pierre-Bénite, France